CLINICAL TRIAL: NCT00507741
Title: Protocol EC-FV-02: A Phase II Study of EC145 in Patients With Advanced Ovarian and Endometrial Cancers
Brief Title: Study of Vintafolide (MK-8109, EC145) in Participants With Advanced Ovarian and Endometrial Cancers (MK-8109-007, EC-FV-02)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8109-007; EC-FV-02 (Other: Endocyte)
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: Cancer; Ovarian; Endometrial; Phase II; EC145; EC20
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Neoplasms | interventions — EC145

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ertafolide + Vintafolide (Experimental): Screening: After completion of all screening procedures and confirmation of eligibility, all participants receive a 1- to 2-mL injection of 0.1 mg ertafolide labeled with 20 to 25 mCi of technetium-99m Part A: Induction phase of treatment: Two 4-week cycles; if stable disease or better at week 8 computed tomography (CT), participant may proceed into maintenance phase, comprised of 4-week cycles with CT every 8 weeks. Participants continue on study until they experience disease progression, unacceptable toxicity, or attain protocol-defined clinical benefit. Part B: 4-week cycles with CT every 8 weeks. Participants continue until they experience disease progression, unacceptable toxicity, or attain protocol-defined clinical benefit.
  Interventions: Drug: Vintafolide; Drug: Ertafolide

INTERVENTIONS:
Drug: Vintafolide — Part A: Induction Phase: vintafolide 1.0 mg intravenous injection, Monday through Friday, for the first 3 weeks of each 4 week cycle. Maintenance Phase: vintafolide 2.5 mg intravenous injection, Monday, Wednesday and Friday, weeks 1 and 3 of each 4 week cycle. At the investigator's discretion, participants may receive vintafolide via an ambulatory pump after the first week of therapy has been administered in the clinic setting. Part B: vintafolide 2.5 mg intravenous injection, Monday, Wednesday and Friday, weeks 1 and 3 of each 4 week cycle. At the investigator's discretion, participants may receive vintafolide via an ambulatory pump after the first week of therapy has been administered in the clinic setting.
Drug: Ertafolide

SUMMARY:
This is a Phase II clinical trial evaluating the benefit from therapy with vintafolide in participants with advanced ovarian and endometrial cancers.

DETAILED DESCRIPTION:
This is a Phase II clinical trial of vintafolide administered to participants with advanced ovarian and endometrial cancers.

Vintafolide is a drug that is specifically designed to enter cancer cells via the folate vitamin receptor (FR). Experimental evidence shows that this target receptor is expressed on virtually all ovarian cancers as well as the majority of endometrial cancers. Early clinical evidence in a small number of Phase I patients suggests that vintafolide may have antitumor effect in women with advanced ovarian cancer and that it is generally well-tolerated. This evidence suggests that vintafolide may be useful as chemotherapy against advanced ovarian and endometrial cancers. The primary objective of Part A of this study is to collect data on clinical benefit produced by therapy with vintafolide. The primary objective of Part B of this study is to collect data on the safety and efficacy of vintafolide.

All participants will undergo imaging with the FR targeting investigational imaging agent ertafolide (EC20, FolateScan) during the screening period to confirm eligibility for the treatment portion of the clinical trial. Clinical evidence suggests that ertafolide may be used to identify women with cancers that express the target receptor.

Information about the safety and tolerability of both vintafolide and ertafolide will be assessed.

ELIGIBILITY:
Part A:

Inclusion Criteria:

* Radiographic evidence of measurable disease (by Response Evaluation Criteria In Solid Tumors [RECIST]) and either:

  * Advanced epithelial ovarian cancer with serous or endometrioid histology, as confirmed by previous biopsy or,
  * ertafolide scan positive ovarian cancer, primary peritoneal cancer or adenocarcinoma of the endometrium.
* Prior treatment with platinum and/or taxane compounds.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2.
* At least 4 weeks from prior therapy and recovered from associated acute toxicities.
* Adequate bone marrow reserve, renal, and hepatic function.
* Negative serum pregnancy test for women of childbearing potential and willingness to practice contraceptive methods.

Exclusion Criteria:

* Serious comorbidities (as determined by the Principal Investigator).
* Women who are pregnant or lactating.
* Symptomatic central nervous system (CNS) metastasis.
* Prior radiation therapy to assessable disease, unless disease progression is confirmed at that site.
* Requires palliative radiotherapy at time of study entry.
* Unable to tolerate conditions for radionuclide imaging.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational.
* Those who have been administered another radiopharmaceutical that would interfere with the assessment of 99mTc-ertafolide scan.

Part B:

Inclusion Criteria:

* Radiographic evidence of measurable disease (by RECIST criteria)
* ertafolide scan positive recurrent or persistent epithelial ovarian, primary fallopian tube, or peritoneal cancer.
* Prior treatment with platinum compounds, but not more than 4 prior cytotoxic chemotheraputic regimens.
* ECOG Performance status of 0-2.
* At least 3 weeks from prior cytotoxic therapy and recovered from associated acute toxicities.
* Adequate bone marrow reserve, renal, and hepatic function.
* Negative serum pregnancy test for women of childbearing potential and willingness to practice contraceptive methods.

Exclusion Criteria:

* Serious comorbidities (as determined by the Principal Investigator).
* Women who are pregnant or lactating.
* Symptomatic CNS metastasis.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational.
* Those who have had prior therapy with Vinorelbine or vinca-containing compounds.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Part A: Percentage of patients deriving clinical benefit. Part B: To gather pilot data on efficacy and toxicity of EC145. | Clinical benefit is defined as the ability to receive 6 or more cycles (i.e., months) of therapy without progression of disease.

SECONDARY OUTCOMES:
Tumor responses to EC145 therapy. | Duration of EC145 therapy will vary according to individual patient response.
Progression-free survival, response duration, and overall survival time observed after EC145 therapy. | 2 years after completing therapy with EC145 and the 30-day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Reddy JA, Dorton R, Westrick E, Dawson A, Smith T, Xu LC, Vetzel M, Kleindl P, Vlahov IR, Leamon CP. Preclinical evaluation of EC145, a folate-vinca alkaloid conjugate. Cancer Res. 2007 May 1;67(9):4434-42. doi: 10.1158/0008-5472.CAN-07-0033. PMID 17483358
- [Derived] Morris RT, Joyrich RN, Naumann RW, Shah NP, Maurer AH, Strauss HW, Uszler JM, Symanowski JT, Ellis PR, Harb WA. Phase II study of treatment of advanced ovarian cancer with folate-receptor-targeted therapeutic (vintafolide) and companion SPECT-based imaging agent (99mTc-etarfolatide). Ann Oncol. 2014 Apr;25(4):852-858. doi: 10.1093/annonc/mdu024. PMID 24667717